CLINICAL TRIAL: NCT03858166
Title: The Efficacy and Safety of Secondary Prophylaxis Versus ANC< 1000/mm3 Administration of PEG-rhG-CSF in Patients Receiving Cytotoxic Chemotherapy for Gynecologic Malignancies
Brief Title: Efficacy and Safety of PEG-rhG-CSF Secondary Prophylaxis vs. Therapeutic Administration in Patients With Ovarian Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Termination
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Beihua Kong, Clinical Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJW-2-PEG-OC
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Adjuvant Chemotherapy; Ovarian Neoplasms; Ovarian Cancer
Keywords: PEG-rhG-CSF; secondary prophylaxis
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): 6mg PEG-rhG-CSF was administrated subcutaneously in 24h after chemotherapy.
  Interventions: Drug: PEG-rhG-CSF
- Adjusted group (Experimental): 6mg PEG-rhG-CSF was administrated subcutaneously when ANC < 1000/mm3 after chemotherapy.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — 6mg PEG-rhG-CSF was administrated subcutaneously at different time after chemotherapy.

SUMMARY:
This study is a multicenter, open-label, randomized clinical trial. Patients with ovarian cancer receiving postoperative adjuvant chemotherapy were eligible to enroll in this study. Eligible patients were randomly allocated in a "1:1" to "Standard group" ( 6mg PEG-rhG-CSF was administrated subcutaneously in 24h after chemotherapy) and "Adjusted group" (6mg PEG-rhG-CSF was administrated subcutaneously when ANC < 1000/mm3 after chemotherapy). All patients need to receive at least 2 cycles of PEG-rhG-CSF administration. The primary outcome is the incidence of grade 3/4 neutropenia, and the duration of grade 3/4 neutropenia, the second outcomes are the incidence of FN, neutropenia-related hospitalization, incidence of reduction and delay of chemotherapy dose and safety of PEG-rhG-CSF.

DETAILED DESCRIPTION:
Patients with ovarian cancer receiving postoperative adjuvant chemotherapy were recruited and randomly allocated in a "1:1" to "Standard group" (6mg PEG-rhG-CSF was administrated subcutaneously in 24h after chemotherapy) and "Adjusted group" (6mg PEG-rhG-CSF was administrated subcutaneously when ANC < 1000/mm3 after chemotherapy). Eligible patients enrolled in this study need to receive 6 cycles of docetaxel or paclitaxel (including liposome paclitaxel) and carboplatin on day 1, every 3 weeks. All patients need to receive at least 2 cycles of PEG-rhG-CSF administration. The primary outcome is the incidence of grade 3/4 neutropenia, and the duration of grade 3/4 neutropenia, the second outcomes are the incidence of FN, neutropenia-related hospitalization, incidence of reduction and delay of chemotherapy dose and safety of PEG-rhG-CSF.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Histopathology or cytology and immunomolecular biology diagnosed with ovarian cancer
3. Grade 3/4 neutropenia appeared in previous chemotherapy
4. accept at least 3 cycles of adjuvant chemotherapy
5. expected survival time ≥ 8 months; KPS>70
6. Normal bone marrow hematopoietic function: ANC≥1.5×109/L, PLT≥80×109/L, Hb≥75g/L, WBC ≥3.0×109/L
7. No obvious abnormalities in electrocardiogram examination, no obvious cardiac dysfunction
8. Liver function: ALT, TBIL, AST <= 2.5 ULN
9. Renal function: Cr, BUN <= 1.5 ULN
10. All patients must agree to take effective contraceptive measures during the study and within 6 months after discontinuing the treatment. Females of childbearing age must be negative in urinary pregnancy test before the treatment.
11. Before the start of the study, all patients have been fully understood the research and the must sign the informed consent.

Exclusion Criteria:

1. Uncontrolled infection, temperature≥38℃
2. patients with bone marrow dysplasia and other hematopoietic dysfunction , or accepted stem cell or bone marrow transplant in 3 months before recruitment
3. undergoing any other clinical trial in 4 weeks before recruitment
4. undergoing radiotherapy in 4 weeks before recruitment
5. Patients with other malignant tumors who have not been cured or have brain metastasis
6. Liver function: ALT, TBIL, AST > 2.5 ULN; If due to liver metastasis, ALT, TBIL, AST > 5 ULN; Renal function: Cr>1.5; Obvious abnormalities in electrocardiogram
7. Severe heart, kidney, liver and other important organs chronic diseases
8. severe and uncontrolled diabetes
9. Pregnancy or lactation in women or women of childbearing age refused to accept contraception
10. People with allergic diseases or allergies, or who are allergic to this or other genetically engineered Escherichia coli-derived biological products
11. Suspected or confirmed drug use, drug abuse, alcoholics
12. Severe mental or neurological disorders affecting informed consent and/or adverse effect presentation or observation
13. HIV positive
14. Syphilis infection
15. The investigator believes that the patient's condition is not suitable for this clinical study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3/4 neutropenia | At the end of cycle 2 (each cycle is 21 days)
  Incidence of grade 3/4 neutropenia
The duration of grade 3/4 neutropenia | At the end of cycle 2 (each cycle is 21 days)
  The duration of grade 3/4 neutropenia

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China